CLINICAL TRIAL: NCT06969313
Title: Telemedicine Intention, Need, Expectations, and Perceived Challenges Among Women With Osteoporosis
Acronym: TINEPCAWO
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Selkin Yılmaz Muluk, specialist physician, Antalya Training and Research Hospital
Other Study IDs: Antalya City Hospital
Record Dates: First submitted 2025-04-28; First posted 2025-05-13 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Osteoporosis; Telemedicine
Keywords: telemedicine; telehealth; patient needs; osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Younger age group: Participants will be divided into two age groups. The younger age group will include participants below 65.
  Interventions: Other: Structured Questionnaire on Telemedicine Needs
- Older age group: Participants will be divided into two age groups. The older age group will include participants equal to or above 65.
  Interventions: Other: Structured Questionnaire on Telemedicine Needs

INTERVENTIONS:
Other: Structured Questionnaire on Telemedicine Needs — Participants will complete a structured questionnaire designed to assess their telemedicine needs, expectations, and current knowledge. The questionnaire includes items on demographics, osteoporosis management, and telemedicine service expectations. No clinical or pharmacological intervention will be applied.
  Other Names: There is no other intervention.

SUMMARY:
This study aims to explore the needs and expectations of women with postmenopausal osteoporosis regarding telemedicine services. Osteoporosis is a common condition among postmenopausal women that increases the risk of fractures and significantly affects quality of life. Many patients do not receive enough information about their disease and treatments during routine clinic visits, which may affect their ability to manage osteoporosis effectively. Participants will be divided into two age groups: those younger than 65 and those aged 65 or older. These subgroups will be compared in terms of their willingness to use telemedicine, their perceived need for such services, their expectations, preferred service topics, and anticipated barriers.

Telemedicine-including video consultations, remote monitoring, and online health education-can offer support to patients, especially for those facing difficulties in accessing healthcare, such as elderly individuals, those living in rural areas, or people with mobility issues.

In this research, women aged 50 to 85 who have been diagnosed with postmenopausal osteoporosis will be asked to complete a survey. The survey includes questions about their needs for telemedicine services, including which types of services (such as medication counseling, exercise programs, dietary advice, psychological support) would be most helpful for them.

The study will also examine if age, education level, past fractures, or family history of osteoporosis influence patients' preferences for telemedicine. By identifying these needs, this research aims to improve access to healthcare and develop personalized telemedicine services for women with osteoporosis in Turkey.

This is a non-interventional, observational, and anonymous survey-based study that will take approximately 10-15 minutes to complete. No medications, treatments, or physical tests will be applied.

DETAILED DESCRIPTION:
This observational, cross-sectional study investigates the actual needs, preferences, and expectations of postmenopausal women with osteoporosis regarding the use of telemedicine services. Osteoporosis is a chronic, progressive condition characterized by decreased bone density and increased fracture risk, which can significantly impair mobility, and overall quality of life. Access to ongoing medical support is crucial for these patients, yet many-particularly older individuals-encounter substantial barriers such as physical limitations, transportation difficulties, limited caregiver availability, or lack of local specialist services.

Telemedicine has gained prominence as a solution to these challenges, offering remote access to healthcare services through technologies like video consultations, telephone check-ins, and online education tools. While telemedicine has been widely implemented during the COVID-19 pandemic, there remains a lack of data on how women with postmenopausal osteoporosis view these services, what features they find most useful, and what obstacles they anticipate.

The primary objective of this study is to evaluate which types of telemedicine services are most needed and preferred by this patient population-for example, support related to medication use, exercise programs, and dietary advice. The study also aims to determine whether specific sociodemographic and clinical variables-such as age, education level, marital status-are associated with participants' willingness to use telemedicine and their actual need for it.

To examine age-related differences, participants will be divided into two subgroups: those under 65 years of age and those aged 65 or older. These subgroups will be compared across multiple domains, including their interest in using telemedicine, actual necessity for such services (calculated according to parameters living alone, not driving/owning a car, having a chronic disease other than osteoporosis), expectations for care delivery, preferred content areas, and potential barriers (such as lack of internet access or digital literacy).

Data will be collected using a structured, self-administered questionnaire developed through expert consultation and adapted from validated tools in previous telehealth research. The questionnaire includes closed-ended questions and will be distributed during routine outpatient visits at two regional hospitals. Participants will be informed about the purpose of the study and assured of full anonymity and confidentiality. Completing the questionnaire is voluntary and is estimated to take approximately 10-15 minutes.

By identifying telemedicine-related needs specific to postmenopausal women with osteoporosis, this study seeks to support the creation of age-appropriate, patient-centered telehealth models. These findings may also inform healthcare providers and policymakers on how to design and implement accessible, effective, and equitable digital healthcare interventions to improve long-term disease management and patient outcomes in this growing patient population.

ELIGIBILITY:
Inclusion Criteria:

Female patients aged 50 to 85 years. Diagnosed with osteoporosis (based on clinical evaluation and prior diagnosis). Able to understand and complete the study questionnaire (adequate cognitive function).

Willing and able to provide informed consent and voluntarily participate in the study.

Exclusion Criteria:

Presence of severe medical conditions that may interfere with participation, including:

Severe cardiac diseases (e.g., advanced heart failure). Severe pulmonary diseases (e.g., advanced chronic obstructive pulmonary disease).

Advanced-stage cancer or other life-limiting illnesses. Cognitive impairment preventing understanding or completion of the questionnaire.

Participation in another clinical or interventional study at the same time. Recent significant trauma (physical or psychological) that may interfere with study participation.

Individuals who cannot understand the study goals and risks, or who refuse informed consent.

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals who self-identify as women and are biologically female are eligible to participate in this study. The study focuses on postmenopausal osteoporosis, a condition that occurs in biological females after menopause. Participants must be women aged 50 to 85 years with a confirmed diagnosis of postmenopausal osteoporosis.
Study Population: The study population will include postmenopausal women aged 50 to 85 years with a confirmed diagnosis of osteoporosis. Participants will be recruited from patients attending the Physical Medicine and Rehabilitation Department of Antalya City Hospital and the Gynecology Department of Antalya Anadolu Hospital. To reduce selection bias, a systematic sampling method was employed, whereby every third consecutive woman with osteoporosis who presented to the outpatient clinics during the data collection period was invited to participate in the study.
Sampling Method: Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Intention to Use Telemedicine Services | Day 1
  Participants were directly asked in the questionnaire about their willingness to use telemedicine services. Response options included "Yes," "Not sure," and "No."
Telemedicine Needs Index | Day 1
  The Telemedicine Need Index was calculated based on three demographic factors: living alone (scored 1), not driving or owning a car (scored 1), and having a chronic disease other than osteoporosis (scored 1). These scores were summed, yielding a total score ranging from 0 to 3. A score of 2 or higher indicated a high need for telemedicine services. Higher scores reflected a greater need for telemedicine.
Differences of telemedicine willingness and need between age groups | Day 1
  Intention to use telemedicine services (answers as yes, not and not sure) and the need for telemedicine (Telemedicine Need Index (scored 0 to 3)) were compared between younger (below 65) older (equal to or above 65) participant.

SECONDARY OUTCOMES:
Patient-reported barriers to telemedicine use | Day 1
  Identification of barriers via questionnaire (technological, privacy, etc.).
Preferred topics for telemedicine services | Day 1
  Patient preferences for telemedicine content (e.g., medication, diet).
Perceived impact of telemedicine on Quality of Life | Day 1
  Likert-scale rating of expected impact of telemedicine on quality of life. Participants rated the perceived impact of telemedicine on their quality of life using a 5-point Likert scale: 1 = Not effective at all, 2 = Slightly effective, 3 = Moderately effective, 4 = Very effective, 5 = Extremely effective. Higher scores indicate a stronger belief that telemedicine services will improve quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Selkin Yilmaz Muluk, MD, Study Chair — Antalya City Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Antalya City Hospital, Antalya
  - Antalya Anatolia Hospital, Antalya

IPD SHARING:
Plan to Share IPD: Yes
IPD related to demographics (such as age and education level, marital status), and responses to the telemedicine needs questionnaire will be available upon reasonable request from the corresponding author. No personally identifiable information will be shared.
Time Frame: IPD will be available from six months after publication to researchers who provide a methodologically sound proposal. Data will be available for a period of one year after publication. Supporting information such as the study protocol and ICF can also be shared upon reasonable request. Data sharing requests should be directed to the corresponding author.
Access Criteria: Access to anonymized IPD and supporting documents will be granted to researchers with a valid scientific proposal that addresses a related research question. Interested researchers must submit a formal request to the corresponding author, including a description of the proposed research, ethical approval (if applicable), and a data use agreement. Data will be shared in anonymized format to protect participant confidentiality.

REFERENCES:
- [Background] Sasaki R, Yunoki T, Nakano Y, Fukui Y, Takemoto M, Morihara R, Abe K, Yamashita T. Actual Telemedicine Needs of Japanese Patients with Neurological Disorders in the COVID-19 Pandemic. Intern Med. 2023 Feb 1;62(3):365-371. doi: 10.2169/internalmedicine.9702-22. Epub 2022 Nov 23. PMID 36418105
- [Background] Palacios S, Neyro JL, Fernandez de Cabo S, Chaves J, Rejas J. Impact of osteoporosis and bone fracture on health-related quality of life in postmenopausal women. Climacteric. 2014 Feb;17(1):60-70. doi: 10.3109/13697137.2013.808182. Epub 2013 Jul 30. PMID 23710562
- [Background] Sood S, Mbarika V, Jugoo S, Dookhy R, Doarn CR, Prakash N, Merrell RC. What is telemedicine? A collection of 104 peer-reviewed perspectives and theoretical underpinnings. Telemed J E Health. 2007 Oct;13(5):573-90. doi: 10.1089/tmj.2006.0073. PMID 17999619